CLINICAL TRIAL: NCT05133024
Title: Use of Beetroot Juice to Protect Against Postoperative Ileus Following Colorectal Surgery: BEET IT Study
Acronym: BEET IT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BC-06366
Record Dates: First submitted 2021-09-27; First posted 2021-11-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Intervention Model Description: Multicentric double-blind randomized controlled prospective phase II study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Beetroot juice bottles are delivered at the central investigational site in labeled boxes indicating whether they are active or control juice. The bottles themselves are identical in appearance and only distinguishable by the manufacturer through the production code. Blinding of the juices is done by an independent party who is responsible for removing the labels, indicating whether the juices are active or nitrate-depleted juice, from the boxes, and assigning an intervention letter code to active or control beetroot juice as 'A' or 'B', without revealing which is which. Sets of 7 bottles, corresponding with the dosage regimen, from A or B according to the randomization list made by an independent statistician, are then labelled with an unique randomization letter code comprising of 2 randomly generated letters, followed by an underscore and a numerical index from 1 to 7 (e.g. AX_1,…, AX_7) to assure allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beetroot juice (Active Comparator): Brand: BEET IT sport NITRATE 400 concentrated beetroot shot (James White Drinks Ltd.) Dosage regimen: 7 shots of 70 mL, once daily in the morning, on 7 consecutive days before surgery
  Interventions: Dietary Supplement: concentrated beetroot juice
- nitrate-depleted beetroot juice (Placebo Comparator): Brand: BEET IT sport NITRATE 400 nitrate-depleted concentrated beetroot shot (James White Drinks Ltd.) Dosage regimen: 7 shots of 70 mL, once daily in the morning, on 7 consecutive days before surgery
  Interventions: Dietary Supplement: concentrated beetroot juice

INTERVENTIONS:
Dietary Supplement: concentrated beetroot juice — Nitrate supplementation; natural source of dietary nitrate
  Other Names: BEET IT sport NITRATE 400 concentrated beetroot shot

SUMMARY:
The goal of the BEET IT study is to examine if preoperative intake of beetroot juice can ameliorate gastrointestinal (GI) recovery after colorectal surgery and thereby help to reduce the duration of postoperative ileus (POI) and prevent prolonged POI. Adult patients undergoing laparoscopic colorectal surgery are randomized 1:1 to consume either concentrated beetroot juice (active intervention) or nitrate-depleted concentrated beetroot juice (placebo) during the week before their surgery. Blood, tissue and/or fecal samples are collected at specific time points pre- and/or postoperatively to study markers related to inflammation, oxidative stress and GI function. Patients are followed from the week before surgery (start of the intervention) until 3 months post-surgery. The study takes place at 5 hospitals in Flanders, Belgium.

DETAILED DESCRIPTION:
Postoperative ileus (POI), a transient impairment of gastrointestinal (GI) motility, remains one of the most common complications following abdominal surgery. It is characterized by the presence of nausea and vomiting, the inability to tolerate oral diet, abdominal distension and delayed passage of flatus and stool. POI usually resolves within 3 to 5 days, but when prolonged, it can lead to increased morbidity, prolonged hospitalization and increased healthcare costs. In patients undergoing colorectal surgery, the reported incidence of prolonged POI (PPOI) is 10.2%. Prevention and treatment remains mainly supportive and no single effective treatment is currently available. Because of its multifactorial origin and possible exogenous factors, prevention and treatment generally requires a multimodal approach. Many of these strategies are part of the Enhanced Recovery after Surgery (ERAS) program. The pathophysiology of POI is marked by an acute neurogenic phase followed by a prolonged inflammatory phase and alterations in the enteric neurotransmission. The pathogenesis involves inflammation and oxidative stress, similar to ischemia/reperfusion (I/R) injury. Both I/R injury and POI are associated with downregulation of nitric oxide (NO) synthases. In this sense, beetroot juice holds considerable promise. Beetroot is a rich source of inorganic nitrate. Consumption of nitrate-rich foods increases the concentration of NO metabolites in the blood and tissues via the enterosalivary nitrate-nitrite-NO pathway, independently of the traditional pathway via the endogenous NOS enzymes, which tends to become less effective in older age and in environments wherein oxygen availability is limited such as during hypoxia and I/R injury. Interest goes to the effects of preoperative beetroot juice supplementation on postoperative GI recovery and POI duration after laparoscopic colorectal surgery. A proof of concept study with 12 patients at our lab already showed promising results. We now want to validate the results in a bigger group of patients via a multicentric double-blind randomized controlled prospective phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective colonic and upper rectum laparoscopic surgery requiring an anastomosis, without the need of conversion

Exclusion Criteria:

General:

* < 18 years of age
* Pregnancy or breast feeding

Medical:

* Psychiatric pathology capable of affecting comprehension and judgment faculty
* History of inflammatory bowel disease
* Chronic vascular disease affecting the intestines
* Chronic constipation (<= 2 bowel movements/week)
* Previous abdominal or pelvic radiation treatment
* Recent (< 3 months before inclusion) or current intra-abdominal infection or inflammation (e.g. diverticulitis, appendicitis, cholecystitis)
* Use of gut motility influencing agents (e.g. tricyclic antidepressants, chronic use of laxatives)
* Use of nitrates (e.g. isosorbide dinitrate, nitroglycerin), including daily consumption of beetroot juice (unless stopped for a month prior to the intervention period)
* Hypotension (< 100/60 mmHg)
* Uncontrolled diabetes mellitus
* Renal or hepatic insufficiency
* Known allergies or intolerances to beetroot, nitrates/nitrites
* Enrollment in other clinical trials/experiments, unless approved by the Ethics Committee(s)

Surgical:

* History of prior colorectal surgery
* Emergency surgery
* Open surgery
* Colorectal surgery not requiring an anastomosis (e.g. colotomy, wedge resection)
* More than 1 bowel anastomosis planned
* Concomitant surgical procedures required (e.g. resection of liver or lung metastases)
* Protective stoma planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery of gastrointestinal (GI) function | hours after the end of surgery (suture)
  composite endpoint requiring recovery of both upper GI functions (tolerance of a solid diet) and lower GI functions (passage of flatus and stool)

SECONDARY OUTCOMES:
First passage of flatus | first occurence after the end of surgery (suture)
  recorded in postoperative days (standard of care) and hours (self-reported in the patient diary)
First passage of stool | first occurence after the end of surgery (suture)
  recorded in postoperative days (standard of care) and hours (self-reported in the patient diary)
First tolerance of liquids | first occurence after the end of surgery (suture)
  liquids: no chewing required, can be quickly swallowed as such, can be ingested with a straw (e.g. water, coffee, tea, juice, soda), recorded in postoperative days (standard of care) and hours (self-reported in the patient diary)
First tolerance of a semi-solid diet | first occurence after the end of surgery (suture)
  semi-solid food: no or limited biting and chewing required, can be easily swallowed, usually ingested with a spoon or fork (e.g. yoghurt, eggs, soft cheeses), recorded in postoperative days (standard of care) and hours (self-reported in the patient diary)
First tolerance of a solid diet | first occurence after the end of surgery (suture)
  solid food: proper and sustained biting and chewing required, cannot be swallowed as such, a knife is usually required to cut the food (e.g. steak, raw vegetables, crisp fruit), recorded in postoperative days (standard of care) and hours (self-reported in the patient diary)
Incidence and recovery of PPOI | until hospital discharge after surgery
  according to the PPOI definition of Vather et al., 2013
Postoperative length of hospital stay | until hospital discharge after surgery
  from the end of surgery (day 0) until discharge (alive) from hospital, recorded in days (standard of care)
Number and types of postoperative complications | until 3 months after surgery
  according to Clavien-Dindo, CCI
Levels of specific biomarkers in blood, tissues and/or feces | 4 time points: (1) inclusion, (2) day of surgery, (3) postoperative day 1, (4) postoperative day 3
  markers for inflammation and oxidative stress, NO bioavailability, intestinal barrier function and permeability

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (6):
  - Antwerp University Hospital, Edegem
  - Hospital East-Limburg, Genk
  - AZ Sint-Lucas Ghent, Ghent
  - Ghent University Hospital, Ghent
  - University Hospital Leuven, Leuven
  - VITAZ, Sint-Niklaas